CLINICAL TRIAL: NCT01641068
Title: Behavioral and Neural Indices of Cognitive Rehabilitation in Women's Cancer: A Pilot Study
Brief Title: Memory and Thinking Skills Workshop to Improve Cognition in Gynecologic and Breast Cancer Survivors With Cognitive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7750; NCI-2012-01035 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7750 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Breast Carcinoma; Cancer Survivor; Cognitive Side Effects of Cancer Therapy; Malignant Female Reproductive System Neoplasm
Keywords: Memory; Attention; Chemo-brain; Survivor; Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (memory and thinking skills workshop) (Experimental): Patients participate in a memory and thinking skills workshop once weekly for 7 weeks. Patients complete cognitive tests and questionnaires at pre-baseline (Visit 1), baseline (Visit 2), and 7 weeks (Visit 3).
  Interventions: Other: Cognitive Intervention; Procedure: Functional Magnetic Resonance Imaging; Other: Memory Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Education Workshop) (Active Comparator): Patients participate in 7 weekly 1-hour group workshops focusing on increasing knowledge and education on the brain and cognition. Patients complete cognitive tests and questionnaires at pre-baseline (Visit 1), baseline (Visit 2), and 7 weeks (Visit 3). Patients are then given the option to participate in the memory and thinking skills workshop.
  Interventions: Other: Educational Intervention; Procedure: Functional Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cognitive Intervention — Participate in memory and thinking skills workshop
  Arms: Arm I (memory and thinking skills workshop)
Other: Educational Intervention — Participate in workshops focusing on increasing knowledge and education on the brain and cognition
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (Education Workshop)
Procedure: Functional Magnetic Resonance Imaging — Undergo functional neuroimaging
  Other Names: fMRI; FUNCTIONAL MRI
Other: Memory Intervention — Participate in memory and thinking skills workshop
  Arms: Arm I (memory and thinking skills workshop)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The purpose of this study is to examine thinking abilities, mood, and quality of life in cancer survivors before and after an 8-week group-based memory and thinking skills workshop. Research participants will include people treated for cancer in the past. Researchers would like to know if there is a relationship between baseline performance on timed attention and memory tasks before receiving memory and thinking skills workshop designed to improve cognition, and performance on such tasks after the workshop.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To objectively assess changes in cognitive performance and quality of life (QOL) pre and post participation in a cognitive rehabilitation intervention in gynecologic and breast cancer survivors who have undergone chemotherapy.

II. To measure changes in neural function as measured by functional magnetic resonance imaging (fMRI) blood oxygenation level dependent (BOLD) signal and corresponding behavioral responses while performing cognitive tasks.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (Skills workshop): Patients participate in a memory and thinking skills workshop once weekly for 7 weeks. Patients complete cognitive tests and questionnaires at pre-baseline (Visit 1), baseline (Visit 2), and 7 weeks (Visit 3).

ARM II (Education workshop): Patients participate in education workshop for 7 weeks 1-hour duration group focusing on the brain and cognition. Patients complete cognitive tests and questionnaires at pre-baseline (Visit 1), baseline (Visit 2), and 7 weeks (Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Subjective concern about declines in cognitive functioning related to a diagnosis of cancer and/or cancer related treatment
* Prior treatment of gynecologic or breast cancer with chemotherapy
* Completion of treatment (e.g., chemotherapy, radiation therapy, surgery, etc.) for gynecologic or breast cancer 6 months or greater in the past
* Able to comprehend and speak English
* For the subset of participants who will undergo magnetic resonance imaging (MRI), ability to withstand lying down in small area (MRI scanner) for 50 minutes
* Completion of successful fMRI safety screening
* Able to give informed consent
* Able to undergo informed consent procedures and 3 hours of testing, plus 8 1-hour cognitive rehabilitation sessions with breaks

Exclusion Criteria:

* Ongoing treatment for ovarian or other cancer (e.g., chemotherapy, radiation, surgery, etc.)
* Cancer onset before the age of 21
* Unstable medical problems (such as unstable heart disease, unstable hypertension, diabetes in poor control, respiratory disease complicated by hypoxia or hypercapnia, infectious illnesses, unstable thyroid dysfunction, currently hospitalized)
* History of, or current symptoms of, serious psychiatric disorder requiring antipsychotic medications or hospitalization; mild depression or stable anti-depressants, and anti-seizure medications are acceptable; anti-anxiety medications may be acceptable
* Current alcohol over-use as defined by currently consuming 4 drinks or more per day or binge drinking (6 or more drinks in one night) within the past week
* History of or current neurological illness that significantly impacts cognition (e.g. stroke, multiple sclerosis, Parkinson's disease, Alzheimer's disease, head injury, epilepsy, etc)
* History of brain injury that significantly impacted cognition; as indicated responses on the Ohio State University Traumatic Brain Injury Identification Method (OSU TBI-ID) greater or equal to any of the following: 30 minutes or more of loss of consciousness (LOC), two or more mild cases within two weeks of each other, or any injury with loss of consciousness before the age of 15
* History of central nervous system (CNS) tumor
* A score of 25 or more on the Patient Health Questionnaire (PHQ-9) on the first visit
* A score of 26 or below on the Mini Mental Status Exam (MMSE) triggers a review by an investigational team before enrolling
* A score above 45 on the Wender Utah Rating Scale for attention deficit disorder (ADD) (WURS)
* For the subset of participants undergoing neuroimaging:

  * Medical history or devices which make an MRI unsafe or uncomfortable (e.g., magnetic rods or pins, metal plates or screws, pacemaker)

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in score on the FACT-Cog-addendum, quality of life (SF-36) questionnaire | Pre-workshop to 7 weeks post-workshop
  Participants respond to questions about their quality of life. The resulting score pre-workshop is compared to the score at 7 weeks post-workshop.
Change in score on the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) questionnaire | Pre-workshop to 7 weeks post-workshop
  Participants respond to questions about their perceived cognitive function. The resulting score pre-workshop is compared to the score at 7 weeks post-workshop.
Changes in neural function measured by fMRI BOLD signal | Pre-workshop to 7 weeks post-workshop
  MRI functional imaging assessments while performing cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Gray, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States